CLINICAL TRIAL: NCT04550585
Title: Specialized Technology Education for Pumps & Pens in Underserved Populations With Diabetes
Acronym: STEPP-UP
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Anne Peters, Professor of Medicine, Clinical Scholar, University of Southern California
Other Study IDs: STEPP-UP
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Type1diabetes
Keywords: low-literacy, diabetes education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Education: Session 1 - Basics of type 1 management — In a group education session, a diabetes educator provides educational session 1 - Basics of type 1 management.
  Accompanying educational guide:
  How Can I Manage My Type 1 Diabetes Better?
Other: Session 2 - Carbohydrate counting — In a group education session, a diabetes educator provides educational session 2 - Carbohydrate counting
  Accompanying educational guide:
  How Can I Manage My Type 1 Diabetes Better?
Other: Education: Session 3 - Insulin self- adjustment — In a group education session, a diabetes educator provides educational session 3 - Insulin self- adjustment
  Accompanying educational guide:
  How Can I Manage My Type 1 Diabetes Better?
Other: Education: Session 4 - Sick day rules and physical activity dose adjustments — In a group education session, a diabetes educator provides educational session 4 - Sick day rules and physical activity dose adjustments
  Accompanying educational guide:
  How Can I Manage My Type 1 Diabetes Better?
Other: Education: Session 5 - Starting the insulin pen (for pen users) or pump (for pump users) — In a group education session, a diabetes educator provides educational session 5 - Starting the insulin pen (for pen users) or pump (for pump users)
  Accompanying educational guide:
  Is the Insulin Pump Right for Me? How Do I Use an Insulin Pump? Is the Insulin Pen Right for Me?
Other: Education: Session 6 - Trouble shooting the pump (for pump users) — In a group education session, a diabetes educator provides educational session 6 - Trouble shooting the pump (for pump users)
  Accompanying educational guide:
  Is the Insulin Pump Right for Me? How Do I Use an Insulin Pump?

SUMMARY:
Lower socioeconomic status (SES) individuals with type 1 diabetes have poorer outcomes than wealthier patients and part of this disparity comes from a lack of tools and knowledge about how to teach these patients on the technologies other patients take for granted. Therefore, this is a study designed to develop and test low literacy English/Spanish language teaching tools for patients with type 1 diabetes treated with varying types of technology in the Los Angeles County healthcare system. The aims are to:To reduce health disparities for underserved adults with diabetes on multiple daily injection (MDI) therapy using vials and syringes through the use of a simplified lower literacy, culturally and language appropriate approach to teach, implement and follow these individuals started on insulin pens and pumps/continuous subcutaneous insulin infusion (CSII); To show no increase in rates of diabetic ketoacidosis (DKA) or severe hypoglycemia when using CSII or pen therapy compared to baseline rates; To reduce time spent in hyper and hypoglycemic ranges, as well as glycemic variability, as measured by blinded continuous glucose monitoring (CGM); Reduce psychological distress due to diabetes and improve health-related quality of life, as measured by validated distress and quality of life scales. Secondary Aims include: Reduction in A1C levels with CSII/pen therapy compared to standard MDI treatment; and to perform a cost-analysis of the process of implementation to improve the generalizability of the model.

DETAILED DESCRIPTION:
SUMMARY OF STUDY RATIONAL - Lower socioeconomic status (SES) individuals with type 1 diabetes (T1D) have poorer outcomes than wealthier patients and part of this disparity comes from a lack of tools and knowledge about how to teach these patients on the technologies other patients take for granted. Until recently many of these lower SES individuals did not have access to health insurance, but with the implementation of the Affordable Care Act the group with the greatest expansion of coverage is the young adult age group (ages 18 - 34), particularly in the Latino community. Increased insurance allows for access to newer technology including insulin pens and pumps. As these patients have not had access to such devices, low literacy educational tool are necessary for safe and efficient utilization. Therefore, this is a study designed to develop and test low literacy English/Spanish language teaching tools for patients with type 1 diabetes treated with varying types of technology in the Los Angeles County (LAC) healthcare system. This study is a single center pilot study and by the nature of our clinic setting it cannot be a randomized controlled trial - it is more of a naturalistic experiment comparing each patient to their prior state of glycemic control with their status after the educational intervention using low-literacy educational materials has been applied.

INTERVENTION - Baseline Visit: Participants will sign informed consent, complete questionnaires, and measure HbA1C. Those opting to do so will start a continuous glucose monitor (CGM) sensor. All patients will be provided the written low literacy teaching tools in the language of their choice.

CGM Visit - for those opting to wear CGM will occur at Week 2 where 14 days of CGM data will be downloaded from participants' device.

Education Sessions: Educational sessions will be conducted using the low-literacy tools we created. Classes will be available on Fridays during T1D Clinic and on Saturdays to maximize participation. Classes will be every two weeks for approximately 3 months. Classes will be approximately 1 ½ hours in duration. Patients will be encouraged but not required to attend the classes. However, those starting on the pen and/or pump will be asked to attend the relevant sessions to prepare them for use of the technology.

Educational Sessions:

Session 1 - Basics of type 1 management Session 2 - Carbohydrate counting, Session 3 - Insulin self- adjustment, Session 4 - Sick day rules and physical activity dose adjustments Session 5 - Starting the insulin pen (for pen users) or pump (for pump users) Session 6 - Trouble shooting the pump (for pump users)

Phone Calls - Each patient will be contacted monthly (baseline month up to month 3 visit) by the diabetes educator to follow-up on questions and concerns regarding their diabetes management.

Clinic Visit 2 - post education visit will occur at 3 months. Questionnaires will be administered, A1C measured and CGM data and compare to baseline.

Clinic Visit 3 - will occur at 6 months. Questionnaires will be administered, A1C measured and CGM data and compare to baseline.

Clinic Visit 4 -will occur at 12 months. Questionnaires will be administered, A1C measured and CGM data and compare to baseline and 6 months.

DATA COLLECTION AND TESTING PROCEDURES (Baseline, 6 months and 12 months) HbA1c - HbA1c will be obtained using the point of care Siemens DCA Vantage Analyzer.

Continuous Glucose Monitoring (CGM)- A commercially available DexCom G5 or Libre device will be provided and a sensor will be inserted. The participant will receive instructions on calibration, insertions, maintenance, use, and removal of the sensor.

T1D REDEEM Diabetes Distress Questionnaire- The T1D REDEEM Diabetes Distress Questionnaire measures several dimensions of stress related to having type 1 diabetes. It consists of the following 7 subscales: Subscale 1 - Powerlessness (5 items); Subscale 2 - Management Distress (4 items); Subscale 3 - Hypoglycemia Distress (4 items); Subscale 4 - Negative Social Perceptions (4 items); Subscale 5 - Eating Distress (3 items); Subscale 6 - Physician Distress (4 items); Subscale 7 - Friend/Family Distress (4 items). Each question has a 6-choice Likert response format. Administration time is approximately 10 minutes.

Hypoglycemia Fear Survey - The Hypoglycemia Fear Survey measures several dimensions of fear of hypoglycemia among adults with type 1 diabetes. It consists of a 10-item Behavior subscale that measured behaviors involved in avoidance and over-treatment of hypoglycemia and a 13-item Worry subscale that measures anxiety and fear surrounding hypoglycemia, each with a 5-choice Likert response format. Administration time is approximately 10 minutes.

Simplified Diabetes Knowledge Test -The Simplified Diabetes Knowledge Test consists of 23 knowledge test items developed by the Michigan Diabetes Research Training Center (MDRTC). These items represent a test of general knowledge of diabetes and are answered in a true/false/don't know format. The psychometric properties provide information regarding the reliability of the various groups of items, as well as a difficulty index (percent of patients who scored this item correctly), and an item to group total correlation for each item. These data can be reported when describing the use of the test. Administration time is approximately 15 minutes.

Assessment of Sever Hypoglycemia and Diabetic Ketoacidosis -The Assessment of Severe Hypoglycemia and Diabetic Ketoacidosis is an interviewer administered survey assessing if the subject had any episodes of severe hypoglycemia and/or diabetic ketoacidosis since their last study visit. Events are recorded to assess frequency, as is type of assistance required to treat the event. Administration time is approximately 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes
2. Age 18 - 75 years old
3. Currently being treated at the T1D clinic in the LAC/USC Healthcare System
4. No use of CSII or insulin pen in the past 6 months
5. No serious illnesses where life expectancy is <1 year
6. Understand the study requirements and agree to comply with all study visits and procedures.
7. Fluent in English or Spanish

Exclusion Criteria:

1. Subject is currently pregnant or lactating or plan on becoming pregnant during the course of the study.
2. Subject is Blind
3. Subject cannot follow instructions due to a medical condition or mental illness.
4. Subject has a known allergy to medical adhesive.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: English or Spanish speaking adults ages 18 to 75 with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Low-literacy based education on HbA1c | 12-months
  Number of patients with decreased HbA1c as measured by point of care HbA1c level from baseline to 12 months
Low-literacy based education on hypoglycemia | 12 months
  Number of patients with decreased hypoglycemia as measured by self report from baseline to 12 months
Low-literacy based education on diabetic ketoacidosis | 12 months
  Number of patients with decreased diabetic ketoacidosis as measured by self report from baseline to 12 months
Low-literacy based education on diabetes distress | 12 months
  Number of patients with decreased diabetes distress as measured by Type 1 Diabetes Reducing Distress and Enhancing Effective Management diabetes distress scale from baseline to 12 months
Low-literacy based education on hypoglycemia fear | 12 months
  Number of patients with decreased hypoglycemia fear as measured by the Hypoglycemia Fear Survey from baseline to 12 months
Low-literacy based education on diabetes knowledge | 12 months
  Number of patients with increased as measured by the Simplified Diabetes Knowledge Test from baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California Eastside Center for Diabetes, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orrange S, Ruelas V, Peters AL. Specialized Technology Education for Pumps and Pens in Underserved Populations with Diabetes. Diabetes Technol Ther. 2022 Apr;24(4):268-275. doi: 10.1089/dia.2021.0265. Epub 2021 Dec 7. PMID 34809482